CLINICAL TRIAL: NCT04855747
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo- Controlled Study to Assess the Efficacy and Safety of REL-1017 as Adjunctive Treatment of Major Depressive Disorder (The RELIANCE-II Study)
Brief Title: A Study to Assess the Efficacy and Safety of REL-1017 as Adjunctive Treatment for Major Depressive Disorder (MDD)
Acronym: RELIANCE-II
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Program Discontinued
Sponsor: Levomecor Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REL-1017-302
Record Dates: First submitted 2021-04-19; First posted 2021-04-22 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-01

CONDITIONS: Major Depressive Disorder; Depression
Keywords: REL-1017; Relmada; NMDA Receptor Antagonist; Esmethadone; Adjunctive; Antidepressant; Reliance; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- REL-1017 25 mg (Experimental): During the double blind treatment period (28 days), participants will take 1 tablet of REL-1017 25 mg, orally, per day in addition to their ongoing antidepressant (ADT)
  Interventions: Drug: REL-1017
- Placebo (Placebo Comparator): During the double blind treatment period (28 days), participants will take 1 tablet of placebo, orally, per day in addition to their ongoing antidepressant (ADT).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: REL-1017 — REL-1017 tablet
  Other Names: Esmethadone
  Arms: REL-1017 25 mg
Drug: Placebo — Placebo tablet
  Arms: Placebo

SUMMARY:
This is an outpatient, 2-arm, Phase 3, multicenter, randomized, double-blind, placebo-controlled study to assess the efficacy and safety of REL-1017 once daily (QD) as an adjunctive treatment of Major Depressive Disorder. Study participants will continue to take their current antidepressant therapy in addition to the study drug or placebo for the duration of the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.0 and 35.0 kg/m2.
* Diagnosed with Major Depressive Disorder (MDD) based on Structured Clinical Interview for DSM-5 (SCID-5) for MDD.
* Current Major Depressive Episode (MDE).
* Treated on approved, stable first-line anti-depressant therapy with inadequate response to 1 to 3 valid courses of treatment with a depressant medication in the current MDE.

Exclusion Criteria:

* Any current and primary psychiatric disorder other than Major Depressive Disorder.
* Severe alcohol or substance use disorder.
* History of bipolar I and II disorder, psychosis, and/or mania.
* Poorly controlled diabetes as defined by HbA1c > 7.5%, despite standard care. Subjects with HbA1c >7.5% may continue in the study if approved by the Relmada Medical Monitor.
* Having received ketamine or esketamine within 60 days prior to Screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-14 (Actual)

PRIMARY OUTCOMES:
Change in the MADRS10 total score | Day 28
  Therapeutic efficacy of REL-1017 as adjunctive treatment versus placebo in the Montgomery-Asberg Depression Rating Scale (MADRS10). A higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6.
  A negative change from baseline indicates improvement.

SECONDARY OUTCOMES:
Change in CGI-S score | Day 28
  Therapeutic efficacy of REL-1017 as an adjunctive treatment versus placebo in Clinical Global Impression of Severity (CGI-S). The CGI-S is a standard method used in clinical studies to quantify and track patient progress and treatment response over time. The scale is composed of 7 ratings: 1 = normal, not at all ill; 2 = borderline ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill patients.
  The score ranges from 1 to 7, and a lower CGI-S score indicates lower levels of depression.
Change in the MADRS10 total score | Day 7
  MADRS10 score at Day 7.
MADRS10 Remission Rate | Day 28
  MADRS10 remission rate (total score ≤10) at Day 28
MADRS10 Response Rater | Day 28
  Improvement ≥50% compared with total Baseline score) at Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Paul Greene, PhD, Study Director — Relmada Therapeutics
Locations (62):
- United States (62):
  - Relmada Site, Homewood, Alabama
  - Relmada Site, Chandler, Arizona
  - Relmada Site, Phoenix, Arizona
  - Relmada Site, Tucson, Arizona
  - Relmada Site, Bryant, Arkansas
  - Relmada Site, Anaheim, California
  - Relmada Site, Bellflower, California
  - Relmada Site, Encino, California
  - Relmada Site, Lafayette, California
  - Relmada Site, Los Angeles, California
  - Relmada Site, Newport Beach, California
  - Relmada Site, Orange, California
  - Relmada Site, Redlands, California
  - Relmada Site, Santa Ana, California
  - Relmada Site, Stanford, California
  - Relmada Site, Temecula, California
  - Relmada Site, Upland, California
  - Relmada Site, Denver, Colorado
  - Relmada Site, Brandon, Florida
  - Relmada Site, Hialeah, Florida
  - Relmada Site, Jacksonville, Florida
  - Relmada Site, Maitland, Florida
  - Relmada Site, Miami, Florida
  - Relmada Site, Miami Springs, Florida
  - Relmada Site, Okeechobee, Florida
  - Relmada Site, Tampa, Florida
  - Relmada Site, West Palm Beach, Florida
  - Relmada Site, Savannah, Georgia
  - Relmada Site, Boise, Idaho
  - Relmada Site, Chicago, Illinois
  - Relmada Site, Elgin, Illinois
  - Relmada Site, Overland Park, Kansas
  - Relmada Site, Marrero, Louisiana
  - Relmada Site, Baltimore, Maryland
  - Relmada Site, Bel Air, Maryland
  - Relmada Site, Gaithersburg, Maryland
  - Relmada Site, Boston, Massachusetts
  - Relmada Site, Bloomfield Hills, Michigan
  - Relmada Site, Mankato, Minnesota
  - Relmada Site, Weldon Spring, Missouri
  - Relmada Site, Las Vegas, Nevada
  - Relmada Site, Toms River, New Jersey
  - Relmada Site, Cedarhurst, New York
  - Relmada Site, Monroe, North Carolina
  - Relmada Site, Beachwood, Ohio
  - Relmada Site, Cincinnati, Ohio
  - Relmada Site, Westlake, Ohio
  - Relmada Site, Philadelphia, Pennsylvania
  - Relmada Site, State College, Pennsylvania
  - Relmada Site, Memphis, Tennessee
  - Relmada Site, Austin, Texas
  - Relmada Site, Beaumont, Texas
  - Relmada Site, Bellaire, Texas
  - Relmada Site, Dallas, Texas
  - Relmada Site, Friendswood, Texas
  - Relmada Site, Houston, Texas
  - Relmada Site, Sherman, Texas
  - Relmada Site, Wichita Falls, Texas
  - Relmada Site, Draper, Utah
  - Relmada Site, Rutland, Vermont
  - Relmada Site, Portsmouth, Virginia
  - Relmada Site, Everett, Washington

REFERENCES:
- See also: Related Info — http://reliancestudies.com